CLINICAL TRIAL: NCT05611879
Title: Efficacy and Safety of Tislelizumab With Platinum Doublet Chemotherapy as Neoadjuvant Therapy for Participants With Initially Unresectable Stage III Non-small Cell Lung Cancer: A Single-arm, Phase II Trial
Brief Title: Neoadjuvant of Tislelizumab Combined With Chemotherapy Followed by Surgery in Unresectable Stage Ⅲ NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21416-0-02
Record Dates: First submitted 2022-11-04; First posted 2022-11-10 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: NSCLC, Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy of Tislelizumab with chemotherapy+surgery (Experimental): Participants will receive neoadjuvant Tislelizumab plus double platinum based chemotherapy for 3 cycles, followed by surgical resection.
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed (Nonsquamous NSCLC) or Paclitaxel/Nab-paclitaxel(Squamous NSCLC); Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab: 200mg, IV, day 1 of each 21-day cycle, Neoadjuvant therapy : 3 cycles
Drug: Pemetrexed (Nonsquamous NSCLC) or Paclitaxel/Nab-paclitaxel(Squamous NSCLC) — Pemetrexed: 500 mg/m^2, IV, day 1 of each 21-day cycle, 3 cycles. Paclitaxel: 60-75mg/m^2, IV, day 1 of each 21-day cycle, 3 cycles. Nab-paclitaxel: 260mg/m^2, IV, day 1 of each 21-day cycle, 3 cycles.
Drug: Carboplatin — AUC 5 mg/mL/min by IV infusion Q3W, given on cycle day 2.

SUMMARY:
The purpose of this conversion therapy study is to evaluate the safety and efficacy of neoadjuvant of Tislelizumab combined with platinum doublet for stage III unresectable locally advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Unresectable stage III non-small cell lung cancer confirmed by histopathology or cytology.
* ECOG score is 0 or 1.
* Adequate hematological function, liver function and renal function.

Exclusion Criteria:

* Previously received systemic anti-tumor therapy for non-small cell lung cancer.
* history or current (non-infectious) pneumonia/interstitial pneumonia requiring steroid treatment.
* History or active pulmonary tuberculosis.
* Active infections that require systemic treatment.
* History or suspected autoimmune disease or immune deficiency who, in the judgment of the investigator, cannot tolerate immunotherapy.
* Untreated active Hepatitis B.
* Has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive).
* Grade 3 or above peripheral neuropathy.
* Severe allergic history to pemetrexed, paclitaxel, albumin-bound paclitaxel, carboplatin or other preventive drugs.
* Underlying severe or uncontrolled disease.
* Malignant tumors other than NSCLC within 5 years.
* Any medical condition requiring systemic treatment with corticosteroids (prednisone or equivalent at a dose of >10mg/ day) or other immunosuppressive agents within 14 days prior to treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Resectability rate | At time of surgery
  Resectability rate is defined as the percentage of patients who were able to undergo surgery after neoadjuvant therapy.

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | At time of surgery
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.
Pathology complete response rate(pCR) | At time of surgery
  pCR rate is defined as the percentage of participants lacking of evidence of viable tumor cells in the pathological examination of resected specimens.
R0 Resection rate | At time of surgery
  R0 Resection rate is defined as the percentage of patients who were able to undergo R0 Resection surgery after neoadjuvant therapy.
Perioperative G3-4 Adverse Events (AEs) | Up to 1 month post surgery
  The number of participants experiencing an perioperative G3-4 AE will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Donghong Chen, Dr., Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No